CLINICAL TRIAL: NCT04889001
Title: Ventilation Knowledge and Skills Retention Among Medical, Nursing and Midwifery Students Using a Novel Tool, the Augmented Infant Resuscitator (AIR) Device as an Instant-feedback Tool / "Electronic Coach".
Brief Title: Ventilation Knowledge and Skills Retention Using a Novel Tool, the Augmented Infant Resuscitator (AIR) Device as an Instant-feedback Tool
Acronym: Sim-II
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mbarara University of Science and Technology (Other)
Collaborators: University of Calgary (Other); The ELMA Foundation (Other); Alberta Children's Hospital Research Institute (Other); Laerdal Foundation (Other); International Development Research Centre, Canada (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020/MUST-4/SIM-II
Record Dates: First submitted 2021-04-30; First posted 2021-05-17 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Ventilation Skills Acquisition and Retention; Ventilation Knowledge Acquisition and Retention

STUDY DESIGN:
Intervention Model Description: Before and after intervention comparison. The students will be trained in simulation enhanced HBB. Simulation enhanced HBB is a one-day course delivered using a format of Explain, Demonstrate and Facilitate practice. Compared to the standard HBB training, the simulation enhanced HBB course is designed with increased peer-to-peer feedback and scripted expert facilitator feedback at HBB practice exercises.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Before/After (Other): Before and after comparison- one arm study
  Interventions: Other: Simulation enhanced HBB training

INTERVENTIONS:
Other: Simulation enhanced HBB training — Simulation enhanced HBB is a one-day course delivered using a format of Explain, Demonstrate and Facilitate practice. Compared to the standard HBB training, the simulation enhanced HBB course is designed with increased peer-to-peer feedback and scripted expert facilitator feedback at HBB practice exercises.

SUMMARY:
Babies born not breathing at birth require effective gentle ventilation to survive and avert organ damage if initial resuscitation steps such as drying, and stimulation are unsuccessful at facilitating breathing. Training of health workers to impart skills on ventilation is a way to prevent these adverse outcomes. Effective ventilation skills are typically acquired through training programs such as Helping Babies Breath (HBB). However, these ventilation skills quickly decay following training and current skills retention methods such as refresher courses are costly and there is a paucity of skilled human resources to effectively facilitate frequent HBB training courses. This raises the need to explore approaches that are independent of retraining for skills maintenance.

The investigators hypothesize that simulation enhanced HBB training followed by self-administered ventilation practice (SAVP) sessions with the Augmented Infant Resuscitator (AIR) as an electronic coach will result into ventilation skills retention over 12 months. SAVP allows participants to maintain practice and training to enhance skills retention.

DETAILED DESCRIPTION:
The investigators will use a multi-methods approach. First, investigators will evaluate the effect of simulation enhanced HBB training and short self-administered practice with AIR device feedback on ventilation skills among undergraduate medical, nursing and midwifery students in Nigeria, Tanzania, and Uganda over a 12-month period. These short practice sessions will be conducted in skills labs. The investigators will equip each skills lab with at least 20 practice stations to enable increased number of students per unit time and reduce total required time in the skills labs for self-practice.

Second, the investigators will conduct focus group discussions with students before and after the intervention, to examine student experiences of simulation with SAVP vis-à-vis their expectations prior and post exposure.

Study design: This will be a 12-month cohort study among medical, nursing and midwifery students rotating in clinical disciplines. We will use a quasi-experimental design and measure ventilation skills before and after administration of a simulation enhanced HBB training plus SAVP with AIR as an intervention. The ventilation skills will also be measured prospectively every 4 months over a 12-month period in HBB scenario settings.

ELIGIBILITY:
Inclusion Criteria:

* Medicine students
* Nursing students
* Midwifery students
* Students at Mbarara University, Busitema University, Lira University, University of Jos

Exclusion Criteria:

* Students outside the participating institutions
* Students outside the Faculty of Medicine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Ventilation skills | 12 months from baseline, after the training program
  Retention of ventilation skills measured using Helping babies breathe Objective Structured Clinical Examinations (OSCE)
Time to effective ventilation | 12 months from baseline, after the training program
  Time in seconds to effective ventilation
Duration of effective ventilation | 12 months from baseline, after the training program
  Time in seconds for the duration of effective ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Data Santorino, MD, Principal Investigator — Mbarara University of Science and Technology

IPD SHARING:
Plan to Share IPD: No
The data involves sensitive information such as video recordings and will therefore not be shared.